CLINICAL TRIAL: NCT04830631
Title: Prediction of Transcranial Direct Current Stimulation (tDCS) Responses Using Electroencephalography (EEG )in Patients With Chronic Stroke
Brief Title: tDCS Response Prediction Using EEG in Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Rusk Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, Won-Seok Kim, Associate professor, Seoul National University Bundang Hospital
Other Study IDs: B-2004/608-004
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Rehabilitation; Transcranial Direct Current Stimulation; Motor Recovery
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cathodal transcranial direct current stimulation (tDCS) over the contralesional motor cortex — Cathodal tDCS will be applied to the contralesional motor cortex with 2mA intesntisy for 30 mins/day. Total 10 sessions will be applied.

SUMMARY:
Patients with chronic stroke (>6 months after stroke) having unilateral upper limb hemiparesis will be recruited. Patients will maintain their usual inpatient rehabilitation including occupational therapy. At baseline (T0) and after 2weeks of enrollment (T1), Fugl-Meyer assessment (FMA) will be assessed at each time. And patients with the changes of FMA between T0 and T1 less than 3 points will be finally recruited. The enrolled patients will receive additional 30-min cathodal transcranial direct current stimulation (tDCS) over the contralesional motor cortex for 10 consecutive weekdays, with maintaining their usual conventional rehabilitation. At T1 and immediately after 10-seessions of tDCS (T2) and 1 month after completing 10-tDCS session (T3), FMA, Actional Research Arm Test (ARAT), Box and Block Test (BBT) and electroencephalography (EEG) were measured.

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 19 to 85 yrs old
* stroke patients with unilateral hemiparesis
* 1st ever stroke
* chronic stroke (>6 months after stroke)

Exclusion Criteria:

* recurrent stroke
* history of traumatic brain injury
* Minimental state examination score is 15 or less.
* Unstable medical conditions
* Severe delirium, disorders of consciousness
* pregnancy
* can not attach tDCS electrode on the scalp due to skin conditions
* can not maintain the sitting position
* intracranial metals

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients with unilateral hemiparesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Fugl-Meyer Assesment Score 1 | Between T1 (before tDCS) and T2 (immediately after completing 10 sessions of tDCS)

SECONDARY OUTCOMES:
Changes in Fugl-Meyer Assesment Score 2 | Between T2 (immediately after completing 10 sessions of tDCS) and T3 (1 month after completing 10 sessions of tDCS)
Changes in Action Research Arm Test Score 1 | Between T1 (before tDCS) and T2 (immediately after completing 10 sessions of tDCS)
Changes in Action Research Arm Test Score 2 | Between T2 (immediately after completing 10 sessions of tDCS) and T3 (1 month after completing 10 sessions of tDCS)
Changes in Box and Block Test Score 1 | Between T1 (before tDCS) and T2 (immediately after completing 10 sessions of tDCS)
Changes in Box and Block Test Score 2 | Between T2 (immediately after completing 10 sessions of tDCS) and T3 (1 month after completing 10 sessions of tDCS)
Changes in EEG index1 | Between T1 (before tDCS) and T2 (immediately after completing 10 sessions of tDCS)
  Various kinds of EEG indexe.g., network indexes, event-related dysynchronization, mu suppression) will be surveyed.
Changes in EEG index 2 | Between T2 (immediately after completing 10 sessions of tDCS) and T3 (1 month after completing 10 sessions of tDCS)
  Various kinds of EEG indexe.g., network indexes, event-related dysynchronization, mu suppression) will be surveyed.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Rusk Rehabilitation Hospital, Seongnam-si, Please Select

IPD SHARING:
Plan to Share IPD: Undecided
After completing the study, EEG indexes and behavioral outcomes will be considered to be shared with researchers who have the clear and reasonable purpose to use our data.